CLINICAL TRIAL: NCT01532089
Title: A Randomized Phase II Trial of Erlotinib Alone or in Combination With Bevacizumab in Patients With Non-Small Cell Lung Cancer and Activating Epidermal Growth Factor Receptor Mutations
Brief Title: Erlotinib Hydrochloride With or Without Bevacizumab in Treating Patients With Stage IV Non-small Cell Lung Cancer With Epidermal Growth Factor Receptor Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC1126; NCI-2012-00053 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-006881; RC1126 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2012-02-07; First posted 2012-02-14 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-07

CONDITIONS: EGFR Exon 19 Deletion Mutation; EGFR NP_005219.2:p.L858R; Lung Non-Squamous Non-Small Cell Carcinoma; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: interventions — Bevacizumab; Immunoglobulin G; Disulfides; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (erlotinib hydrochloride) (Active Comparator): Patients receive erlotinib hydrochloride PO QD on days 1-21. (erlotinib will no longer be supplied and all patients will be removed from study treatment. No further follow-up by any study participants as of September 1, 2019)
  Interventions: Drug: Erlotinib; Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis
- Arm B (erlotinib hydrochloride, bevacizumab) (Experimental): Patients receive erlotinib hydrochloride as in Arm A and bevacizumab IV over 30-90 minutes on day 1. (erlotinib will no longer be supplied and all patients will be removed from study treatment. No further follow-up by any study participants as of September 1, 2019)
  Interventions: Biological: Bevacizumab; Drug: Erlotinib; Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501
  Arms: Arm B (erlotinib hydrochloride, bevacizumab)
Drug: Erlotinib — Given PO
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well erlotinib hydrochloride (Tarceva) with or without bevacizumab (Avastin) works in treating patients with stage IV non-small cell lung cancer (NSCLC) with epidermal growth factor receptor (EGFR) mutations. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, may block tumor growth in different ways by targeting certain cells. Bevacizumab may also stop the growth of NSCLC by blocking the growth of new blood vessels necessary for tumor growth. It is not yet known whether erlotinib hydrochloride is more effective when given alone or with bevacizumab in treating patients with NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the progression-free survival of erlotinib (erlotinib hydrochloride) and bevacizumab versus that of erlotinib alone for the purpose of deciding if the combination arm is worth pursuing in a phase III trial.

SECONDARY OBJECTIVES:

I. To investigate the overall survival of erlotinib and bevacizumab versus erlotinib alone.

II. To investigate the response rate of erlotinib and bevacizumab versus erlotinib alone.

III. To investigate the progression-free survival in patients with exon deletion 19 or exon 21 L858R point mutations.

IV. To investigate the toxicity of erlotinib and bevacizumab versus erlotinib alone using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

CORRELATIVE RESEARCH OBJECTIVES:

I. To correlate EGFR mutations detected in plasma deoxyribonucleic acid (DNA) with those detected in tumor DNA.

II. To estimate the prevalence of EGFR T790M resistance mutations from pretreatment tumor biopsies using more sensitive mutation detection methods.

III. To investigate progression free survival of EGFR mutant NSCLC patients with and without concurrent EGFR T790M detected from pre-treatment tumor specimen using allele specific quantitative polymerase chain reaction (PCR).

IV. To prospectively evaluate the predictive value of plasma VEGF-A levels on progression free survival in patients treated with erlotinib alone or in combination with bevacizumab.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive erlotinib hydrochloride orally (PO) once daily (QD) on days 1-21. (erlotinib will no longer be supplied and all patients will be removed from study treatment. No further follow-up by any study participants as of September 1, 2019)

ARM B: Patients receive erlotinib hydrochloride as in Arm A and bevacizumab intravenously (IV) over 30-90 minutes on day 1. (erlotinib will no longer be supplied and all patients will be removed from study treatment. No further follow-up by any study participants as of September 1, 2019)

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of primary lung carcinoma, non-squamous histology with activating epidermal growth factor receptor (defined as deletion 19 or exon 21 L858R mutation); Note: EGFR mutation testing must be performed at a Clinical Laboratory Improvement Amendments (CLIA) certified lab; either institutional or through a commercial laboratory (e.g. Genzyme, Response Genetics, etc); the laboratory report from the commercial laboratories report the specific mutations detected, and the method of detecting the exon 19 and exon 21 L858R point mutations must be available
* Stage IV disease according to the 7th Edition of the American Joint Committee on Cancer staging system
* Measurable disease
* Life expectancy of >= 12 months
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count (ANC) >= 1,500/mm^3 obtained =< 14 days prior to randomization
* Platelet count >= 100,000/mm^3 obtained =< 14 days prior to randomization
* Hemoglobin >= 9.0 g/dL obtained =< 14 days prior to randomization
* Total bilirubin =< 1.5 x upper limit of normal (ULN) obtained =< 14 days prior to randomization
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x ULN in patients without liver or bone metastases; < 5 x ULN in patients with liver or bone metastases obtained =< 14 days prior to randomization
* Cockcroft-Gault calculated creatinine clearance of >= 45 ml/min or creatinine =< 1.5 x ULN obtained =< 14 days prior to randomization
* Urine dipstick proteinuria < 2+ or urine protein/creatinine (UPC) ratio =< 1.0 obtained =< 14 days prior to randomization

  * Note: patients discovered to have >= 2 + proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate =< 1 g of protein in 24 hours
* Negative pregnancy test done =< 7 days prior to randomization, for women of childbearing potential only
* Provide informed written consent
* Willing to return to Academic and Community Cancer Research United (ACCRU) enrolling institution for follow-up
* Willing to provide tissue and blood samples for correlative research purposes

Exclusion Criteria:

* Mixed, non-small cell and small cell tumors or mixed adenosquamous carcinomas with a predominant squamous component
* Prior chemotherapy or treatment for metastatic non-small cell lung cancer
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive, per medical doctor (MD) discretion
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations, or any other medical condition that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to randomization; EXCEPTIONS: non melanotic skin cancer or carcinoma-in-situ of the cervix; Note: if there is a history of prior malignancy, they must not be receiving other specific treatment (i.e. hormonal therapy) for their cancer
* History of myocardial infarction or other evidence of arterial thrombotic disease (angina), symptomatic congestive heart failure (New York Heart Association >= grade 2), unstable angina pectoris, or cardiac arrhythmia; Note: allowed only if patient has no evidence of active disease for at least 6 months prior to randomization
* History of cerebral vascular accident (CVA) or transient ischemic attack (TIA) =< 6 months prior to randomization
* History of bleeding diathesis or coagulopathy
* Inadequately controlled hypertension (systolic blood pressure of > 150 mmHg or diastolic pressure > 100 mmHg on anti-hypertensive medications); Note: history of hypertensive crisis or hypertensive encephalopathy not allowed
* Current or recent (=< 10 days prior to randomization) use of aspirin (> 325 mg/day), clopidogrel (> 75 mg/day), or prasugrel (> 10 mg/day)
* Serious non-healing wound, ulcer, bone fracture, or have undergone a major surgical procedure, open biopsy, or significant traumatic injury =< 28 days or core biopsy =< 7 days prior to randomization
* History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess =< 6 months prior to randomization
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of hemoptysis >= grade 2 (defined as bright red blood of at least 2.5 mL) =< 3 months prior to randomization
* Known central nervous system (CNS) disease, except for treated brain metastasis; Note: treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS); gamma knife, linear accelerator (LINAC), or equivalent or a combination as deemed appropriate by the treating physician; patients with CNS metastases treated by neurosurgical resection or brain biopsy performed =< 3 months prior to randomization will be excluded; Note: craniotomy or intracranial biopsy site must be adequately healed, free of drainage or cellulitis, and the underlying cranioplasty must appear intact at the time of randomization; study treatment should be initiated > 28 days following the last surgical procedure (including biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity)
* Significant vascular disease (e.g. aortic aneurysm surgical repair or recent peripheral arterial thrombosis) =< 6 months prior to randomization
* Radiotherapy to any site for any reason =< 14 days prior to randomization
* Receiving any medications or substances that are strong or moderate inhibitors of CYP3A4; use of the following strong or moderate inhibitors are prohibited =< 7 days prior to randomization:

  * Strong inhibitors of CYP3A4: indinavir (Crixivan), nelfinavir (Viracept), atazanavir (Reyataz), ritonavir (Norvir), clarithromycin (Biaxin, Biaxin XL), itraconazole (Sporanox), ketoconazole (Nizoral), nefazodone (Serzone), saquinavir (Fortovase, Invirase), telithromycin (Ketek)
  * Moderate inhibitors of CYP3A4: aprepitant (Emend), erythromycin (Erythrocin, E.E.S, Ery-Tab, Eryc, EryPed, PCE, fluconazole (Diflucan), grapefruit juice, verapamil (Calan, Calan SR, Covera-HS, Isoptin SR, Verelan, Verelan PM), diltiazem (Cardizem, Cardizem CD, Cardizem LA, Cardizem SR, Cartia XT, Dilacor XR, Diltia XT, Taztia XT, Tiazac)
* Receiving any medications or substances that are strong or moderate inducers of CYP3A4; use of the following inducers are prohibited =< 7 days prior to randomization: efavirenz (Sustiva), nevirapine (Viramune), carbamazepine (Carbatrol, Epitol, Equetro, Tegretol, Tegretol-XR), modafinil (Provigil), phenobarbital (Luminal), phenytoin (Dilantin, Phenytek), pioglitazone (Actos), rifabutin (Mycobutin), rifampin (Rifadin), St. John?s wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-03-16 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2020-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Stinchcombe, Principal Investigator — Academic and Community Cancer Research United
Locations (19):
- United States (19):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Carle Cancer Center NCI Community Oncology Research Program, Urbana, Illinois
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin

REFERENCES:
- [Derived] Stinchcombe TE, Janne PA, Wang X, Bertino EM, Weiss J, Bazhenova L, Gu L, Lau C, Paweletz C, Jaslowski A, Gerstner GJ, Baggstrom MQ, Graziano S, Bearden J 3rd, Vokes EE. Effect of Erlotinib Plus Bevacizumab vs Erlotinib Alone on Progression-Free Survival in Patients With Advanced EGFR-Mutant Non-Small Cell Lung Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2019 Oct 1;5(10):1448-1455. doi: 10.1001/jamaoncol.2019.1847. PMID 31393548

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Erlotinib Hydrochloride): Patients receive 150 mg erlotinib hydrochloride PO QD on days 1-21.
- Arm B (Erlotinib Hydrochloride, Bevacizumab): Patients receive 150 mg erlotinib hydrochloride as in Arm A and 15 mg/kg bevacizumab IV over 30-90 minutes on day 1.
Period: Overall Study
Arm/Group | Arm A (Erlotinib Hydrochloride) | Arm B (Erlotinib Hydrochloride, Bevacizumab)
Started (Randomized) | 45 | 43
Completed | 45 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Erlotinib Hydrochloride) | Arm B (Erlotinib Hydrochloride, Bevacizumab) | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Continuous [Median (Full Range); unit: years] | 63 [47 to 84] | 65 [31 to 84] | 63.5 [31 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 39 | 36 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 19 | 24 | 43
    1 | 26 | 19 | 45
EGFR exon mutation [Count of Participants; unit: Participants] — Epidermal growth factor receptor (EGFR) exon mutation
  Participants
    Exon 19 deletion | 30 | 29 | 59
    Exon 21 L858R mutation | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as at least a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Time from randomization to disease progression and death of any cause, whichever comes first, assessed up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Erlotinib Hydrochloride) | Arm B (Erlotinib Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 45 | 43
months | 13.5 [8.8 to 21.6] | 17.9 [13.3 to 24.1]
Statistical Analysis 1: Comparison: Arm A (Erlotinib Hydrochloride) vs Arm B (Erlotinib Hydrochloride, Bevacizumab); Test type: Superiority; p = 0.39, Log Rank; Comparisons of PFS between arms were conducted using a stratified log-rank test; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.50 to 1.31]

2. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from randomization to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Time from randomization to death of any causes, assessed up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Erlotinib Hydrochloride) | Arm B (Erlotinib Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 45 | 43
months | 50.6 [49.4 to NA] — The 95% CI upper limit was not reached (insufficient number of participants with events). | 32.4 [26.9 to 54.4]
Statistical Analysis 1: Comparison: Arm A (Erlotinib Hydrochloride) vs Arm B (Erlotinib Hydrochloride, Bevacizumab); Test type: Superiority; p = 0.33, Log Rank; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.71 to 2.81]

3. Secondary Outcome: Response Rate (Complete or Partial) to Each Treatment, Evaluated Using the New International Criteria Proposed by the Revised Response Evaluation Criteria in Solid Tumors Guidelines (Version 1.1)
Description: The response rate (percentage) is the percent of patients whose best response was Complete Response (CR) or Partial Response (PR) as defined by RECIST 1.1 criteria. Percentage of successes will be estimated by 100 times the number of successes divided by the total number of evaluable patients. (CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites).
Time Frame: Up to 6 years
Population: Patients with tumor response data available were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Erlotinib Hydrochloride) | Arm B (Erlotinib Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 42 | 43
percentage of patients | 83 [69 to 93] | 81 [67 to 92]
Statistical Analysis 1: Comparison: Arm A (Erlotinib Hydrochloride) vs Arm B (Erlotinib Hydrochloride, Bevacizumab); Test type: Superiority; p = 0.81, Chi-squared

4. Secondary Outcome: Progression Free Survival of Patients With Different Mutation Types (Exon Deletion 19 Versus Exon 21 L858R)
Description: Progression free survival (PFS) is defined as the time from the date of randomization to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as at least a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator by mutation type.
Time Frame: From the date of randomization to the date of disease progression or death of any cause, whichever comes first, assessed up to 6 years
Population: This analysis includes all patients with EGFR exon mutation data available and primary endpoint data available.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Exon 19 Deletion: Patients with exon 19 deletion EGFR exon mutation.
- Exon 21 L858R: Patients with exon 21 L858R EGFR exon mutation.
Arm/Group | Exon 19 Deletion | Exon 21 L858R
Number analyzed (Participants) | 59 | 29
months | 17.9 [13.5 to 23.9] | 12.6 [9.0 to 24.1]

5. Secondary Outcome: Number of Patients Experiencing Toxicity
Description: The number of patients experiencing toxicity defined as grade 3 or higher adverse events (using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0) considered at least possibly related to treatment is reported below.
Time Frame: Up to 42 days after treatment discontinuation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Erlotinib Hydrochloride) | Arm B (Erlotinib Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 45 | 43
Participants | 13 | 31

6. Other Pre Specified Outcome: EGFR Mutations Detected in Plasma Deoxyribonucleic Acid (DNA)
Description: Agreement of EGFR mutations detected in plasma DNA with those detected in tumor DNA will be evaluated.
Time Frame: Up to 6 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: EGFR Mutations Detected in Tumor Deoxyribonucleic Acid (DNA)
Description: Agreement of EGFR mutations detected in plasma DNA with those detected in tumor DNA will be evaluated.
Time Frame: Up to 6 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Prevalence of EGFR T790M Resistance Mutations From Pretreatment > Tumor Biopsies Using More Sensitive Mutation Detection Methods
Description: Tested using Cox proportional hazard model after adjusting for treatment effect. The robustness of treatment effect in different subgroups will be examined in a Forest plot.
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: EGFR T790M Mutations
Description: Detected from pre-treatment tumor specimen using allele specific quantitative polymerase chain reaction (PCR). The PFS of patients with EGFR T790M mutations will be estimated and the survival difference will be tested using Cox proportional hazard model after adjusting for treatment effect. The robustness of treatment effect in different subgroups will be examined in a Forest plot.
Time Frame: Up to 6 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Predictive Value of Plasma VEGF-A Levels on Progression Free Survival in Patients Treated With Erlotinib Hydrochloride Alone or in Combination With Bevacizumab
Description: Evaluated using time-dependent receiver operating characteristic curve and area under curve.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 42 days after treatment discontinuation
Arm/Group | Arm A (Erlotinib Hydrochloride) | Arm B (Erlotinib Hydrochloride, Bevacizumab)
All-Cause Mortality (participants affected / at risk) | 23/45 | 27/43
Serious Adverse Events (participants affected / at risk) | 12/45 | 17/43
Other Adverse Events (participants affected / at risk) | 43/45 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Erlotinib Hydrochloride) (N=45) | Arm B (Erlotinib Hydrochloride, Bevacizumab) (N=43)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Sudden death NOS (General disorders) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (3) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 4 (4) | 2 (3)
Thromboembolic event (Vascular disorders) | 2 (2) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Erlotinib Hydrochloride) (N=45) | Arm B (Erlotinib Hydrochloride, Bevacizumab) (N=43)
Anemia (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (5)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (4) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (29)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 2 (3) | 2 (5)
Periorbital edema (Eye disorders) | 1 (1) | 1 (2)
Watering eyes (Eye disorders) | 1 (7) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (5)
Anal hemorrhage (Gastrointestinal disorders) | 3 (16) | 3 (24)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 37 (606) | 38 (528)
Dyspepsia (Gastrointestinal disorders) | 1 (4) | 1 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (45)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (10) | 5 (9)
Oral hemorrhage (Gastrointestinal disorders) | 2 (28) | 5 (9)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (28)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (2)
Fatigue (General disorders) | 10 (44) | 14 (39)
Fever (General disorders) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (11) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (5)
Pain (General disorders) | 2 (3) | 1 (1)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (2)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 3 (3)
Nail infection (Infections and infestations) | 2 (5) | 1 (23)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (5)
Paronychia (Infections and infestations) | 6 (37) | 3 (10)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (3) | 1 (2)
Urinary tract infection (Infections and infestations) | 3 (4) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Activated partial throm time prolonged (Investigations) | 1 (9) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (4) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 8 (19) | 1 (4)
Cardiac troponin I increased (Investigations) | 1 (21) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 2 (6)
Lymphocyte count decreased (Investigations) | 5 (33) | 1 (1)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 4 (19) | 6 (33)
Anorexia (Metabolism and nutrition disorders) | 4 (24) | 7 (14)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (20)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 2 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (8) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (4)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (7) | 3 (23)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (3)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (6)
Insomnia (Psychiatric disorders) | 4 (19) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (4)
Hematuria (Renal and urinary disorders) | 15 (102) | 12 (79)
Proteinuria (Renal and urinary disorders) | 15 (106) | 24 (218)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (4)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (8) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (34)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (11) | 3 (54)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (34) | 6 (74)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (17)
Rash acneiform (Skin and subcutaneous tissue disorders) | 40 (586) | 42 (732)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (7) | 3 (11)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 23 (413) | 36 (617)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT01532089/Prot_SAP_000.pdf